CLINICAL TRIAL: NCT03388164
Title: Adherence to Antidepressant Treatment in Subjects With Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early based on the planned interim analysis that did not meet criteria for continuation.
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017-007
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2020-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Escitalopram + RT2CK17 (Active Comparator): 10mg escitalopram + 5mg RT2CK17 will be given orally and encapsulated into one capsule, once per day for 8 weeks. The capsules will be produced in the same manner as the placebo comparator by a local compounding pharmacy in Tulsa, Oklahoma.
  Interventions: Drug: Escitalopram + RT2CK17
- Escitalopram + Placebo (Placebo Comparator): 10mg escitalopram + 5mg placebo will be given orally and encapsulated into one capsule, once per day for 8 weeks. The capsules will be produced in the same manner as the active comparator by a local compounding pharmacy in Tulsa, Oklahoma.
  Interventions: Drug: Escitalopram + Placebo

INTERVENTIONS:
Drug: Escitalopram + RT2CK17 — Participants randomized to active or placebo condition will be prescribed medication over the course of 8 weeks, with in-person follow-up visits at weeks 0, 2, 4 and 8, with follow-up phone calls on weeks 1, 3 and 6.
  Arms: Escitalopram + RT2CK17
Drug: Escitalopram + Placebo — Participants randomized to active or placebo condition will be prescribed medication over the course of 8 weeks, with in-person follow-up visits at weeks 0, 2, 4 and 8, with follow-up phone calls on weeks 1, 3 and 6.
  Arms: Escitalopram + Placebo

SUMMARY:
This study aims to determine whether a combination a first-line antidepressant plus "RT2CK17" in a capsule relative to a first-line antidepressant plus placebo in a capsule results in higher rates of medication adherence in individuals with moderate to severe depression. In this double-blind randomized placebo controlled trial, 100 individuals with a Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) scale score ≥ 14 will be enrolled to participate in an 8 week treatment study. Participants will be randomized with a 1-1 ratio to receive 5 milligrams (mg) "RT2CK17" + 10 mg escitalopram or placebo + 10 mg escitalopram to be taken orally once per day. Participants will undergo a 3 hour baseline evaluation visit at week 0, two 30-minute office visits (week 2 and 4), one 60-minute office visit (week 8) and three 5-minute phone calls (weeks 1, 3, and 6) during which clinical assessments and measures will be obtained. The trial is designed with two stages: 20 participants in Stage 1 will be used to estimate the adherence effect size; Stage 2 is designed with an interim analysis to test our hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Baseline QIDS-SR ≥ 14 (moderate depression)
* Age 18 - 65
* Written Informed Consent
* Major Depressive Disorder, single-episode/recurrent, not in remission

Exclusion Criteria:

* RT2CK17-related exclusions
* Uncontrolled hyperthyroidism
* Glaucoma
* Motor tics
* Monoamine oxidase inhibitor treatment
* Serious coronary artery disease, cardiomyopathy, serious cardiac arrhythmias
* Uncontrolled hypertension
* Peripheral vasculopathy
* Pregnancy
* Bipolar Disorder
* Psychotic Disorder
* History of intolerability of study medications
* Currently taking psychiatric medications
* Current Substance Use Disorder (other than nicotine)
* Current Alcohol Use Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Paulus, M.D., Study Director — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paulus MP, Kuplicki R, Victor TA, Yeh HW, Khalsa SS. Methylphenidate augmentation of escitalopram to enhance adherence to antidepressant treatment: a pilot randomized controlled trial. BMC Psychiatry. 2021 Nov 19;21(1):582. doi: 10.1186/s12888-021-03583-7. PMID 34798853

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three individuals were excluded prior to group assignment:
  2- did not meet inclusion criteria (alcohol use, low TSH)
  1- declined to participate
Period: Overall Study
Arm/Group | Escitalopram + RT2CK17 | Escitalopram + Placebo
Started | 10 | 10
Completed | 7 | 9
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram + RT2CK17 | Escitalopram + Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (10.7) | 31.0 (10.6) | 31.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adherence
Description: To determine whether RT2CK17 + escitalopram results in higher rates of medication adherence relative to placebo + escitalopram as measured by percentage pill count
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Arm/Group | Escitalopram + RT2CK17 | Escitalopram + Placebo
Number analyzed (Participants) | 7 | 9
percentage of pills taken | 93.5 (7.6) | 97.6 (6.5)

2. Secondary Outcome: Adherence Consistency
Description: To determine whether RT2CK17 + escitalopram results in greater consistency of adherence relative to placebo + escitalopram as measured by percentage of doses taken on schedule within 25% of the expected time interval, defined as +/- 6 hours from the participant's breakfast time
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of pills taken on time
Arm/Group | Escitalopram + RT2CK17 | Escitalopram + Placebo
Number analyzed (Participants) | 7 | 9
percentage of pills taken on time | 89.8 (8.2) | 93.6 (8.4)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Escitalopram + RT2CK17 | Escitalopram + Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The study was terminated early based on the planned interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03388164/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT03388164/ICF_001.pdf